CLINICAL TRIAL: NCT07228845
Title: Effectiveness Comparison of 3D-Printed and Conventional Ear Tip Comfort in Individuals With Hearing Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Bryan Wong, Assistant Professor of Practice, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5737
Record Dates: First submitted 2025-11-07; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Hearing Aids; Hearing Loss, Bilateral Sensorineural; 3D Printing
Keywords: hearing aids; 3D printing; hearing loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- In-house Study group_Resin (Experimental): participants will initially receive ear tips fabricated using biocompatible resin
  Interventions: Device: BTE hearing aids with compatible ear tips (Resin, Third-party, FlexRes)
- Third-party Manufactured (Active Comparator): participants will initially receive ear tips fabricated by third party manufacturer using biocompatible resin
  Interventions: Device: BTE hearing aids with compatible ear tips (Third-party, FlexResin, Resin)
- In-house Study group_FlexibleResin (Experimental): Participants will initially receive ear tips fabricated using biocompatible flexible resin
  Interventions: Device: BTE hearing aids with compatible ear tips (FlexResin, Resin, Third-party, FlexResin)

INTERVENTIONS:
Device: BTE hearing aids with compatible ear tips (Third-party, FlexResin, Resin) — Hearing aids will be fit with three different types of customized ear tips. They will wear each ear tip for 1 week. The following order participants will wear each ear tip includes: Third-party, FlexResin, Resin. Hearing aids will be programmed to fit the participants' hearing loss from 250-8000Hz. A short washout period will follow completion of testing with ear tip group.
  Arms: Third-party Manufactured
Device: BTE hearing aids with compatible ear tips (FlexResin, Resin, Third-party, FlexResin) — Hearing aids will be fit with three different types of customized ear tips. They will wear each ear tip for 1 week. The following order participants will wear each ear tip includes: Resin, Third-party, FlexResin. Hearing aids will be programmed to fit the participants' hearing loss from 250-8000Hz. A short washout period will follow completion of testing with ear tip group
  Arms: In-house Study group_FlexibleResin
Device: BTE hearing aids with compatible ear tips (Resin, Third-party, FlexRes) — Hearing aids will be fit with three different types of customized ear tips. They will wear each ear tip for 1 week. The following order participants will wear each ear tip includes: Resin, Third-party, FlexResin. Hearing aids will be programmed to fit the participants' hearing loss from 250-8000Hz. A short washout period will follow completion of testing with ear tip group
  Arms: In-house Study group_Resin

SUMMARY:
Access to affordable and timely hearing healthcare remains a major challenge for many individuals, partly due to the high cost and long turnaround time. This study will explore whether 3D-printed ear tips perform as well as or better than standard ear tips in terms of sound quality, comfort, and fit over a prolonged duration in a sample of individuals with bilateral hearing loss. It will also compare how long each method takes to make and how much each costs.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral, symmetric, sensorineural hearing loss, with thresholds between normal and severe degree of hearing loss
* Normal otoscopy: patent ear canals with normal appearing eardrums and aerated middle ear, bilaterally.
* English speaking.

Exclusion Criteria:

* Self reported history of extensive or current outer or middle ear pathology.
* Self reported history of extensive outer or middle ear surgery.
* Self reported history of neurological or cognitive disorder.
* Active ear infection

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Outer EAR comfort questionnaire | through study completion, an average of 1 week
  A validated questionnaire, Outer EAR, will be used to elicit patient perception of physical comfort, acoustic comfort, quality of voice, and overall self-perceived satisfaction. Includes 6 items (5 levels) , with 5 representing best possible function/rating.
Real Ear Measures | through study completion, an average of 1 week
  Evaluation of ear canal acoustics with participant wearing a hearing aid and eartip type (3d party, in-house_Resin, in-house_FlexResin). A thin microphone tube is placed in the ear canal to measure the average amount gain (dB SPL) across various frequencies (250-8000Hz) while the participant sits in front of a speaker playing sound samples. Results are recorded in gain (dB SPL) across frequencies.

SECONDARY OUTCOMES:
Cost | through study completion, an average of week
  The total raw cost ($, dollars US)
Time | through study completion, an average of week
  Time-to-subject for each ear tip type

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Arizona Hearing Clinic, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No